CLINICAL TRIAL: NCT03361930
Title: Electromyographic Comparison of Muscle Activity in Children With Spastic Unilateral Cerebral Palsy During Walking With Two Different Types of Hinged Ankle-foot Orthoses
Brief Title: Changes in Muscle Activity of Children With Spastic Unilat Cerebral Palsy Using 2 Types of Ankle-foot Orthoses to Walk
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: NITO, Norwegian engineering and technology organiziation (Unknown); Sophies Minde Ortopedi (Industry)
Responsible Party: Principal Investigator, Ann-Britt Huse, Principal investigator, Oslo University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017/161
Record Dates: First submitted 2017-11-16; First posted 2017-12-05 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-11

CONDITIONS: Cerebral Palsy, Spastic; Hemiplegic Cerebral Palsy
Keywords: spastic unilateral cerebral palsy, ankle-foot orthosis, AFO, muscle activity, muscular activity, electromyography, EMG,
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CP participants (Experimental): Single-day data collection for walking conditions; barefoot, with plain ankle-foot orthosis (flat foot plate) on involved side, with tone-reducing ankle-foot orthosis on involved side.
  Interventions: Device: Ankle-foot orthosis

INTERVENTIONS:
Device: Ankle-foot orthosis — Two custom ankle-foot orthoses for the involved lower leg; cast, rectified and fitted by same certified orthotist to reduce clinician variability.
  The cast is rectified according to the specifications of Hylton (1987) to produce tone-reducing features in the foot plate; the tone-reducing ankle-foot orthosis is manufactured on this cast. The orthotist then remodels the cast with a flat foot plate; the plain ankle-foot orthosis is then manufactured.
  Other Names: AFO

SUMMARY:
The aim of this study is to investigate if ankle-foot orthoses affect changes in muscle activity of children with spastic unilateral cerebral palsy during walking.

To minimize investigator variability, the same orthotist CO, clinical gait analyst GA and physiotherapist PT will perform their designated functions for all participants.

Each subject will be required to attend three appointments.

First appointment: CO takes a lower leg cast of the involved side; the cast is taken with the ankle and hindfoot corrected to neutral position.

Second appointment: CO fits the tone-reducing ankle-foot orthosis which entails trimming the device to fit footwear, checking the orthotic device restricts plantarflexion and ensuring comfortable and functional fit. The device is modified with holes for electrode placement at locations for tibialis anterior and gastrocnemius identified by PT.

The child receives the tone-reducing ankle-foot orthosis and is instructed to use this orthotic device on a daily basis for the next four weeks to grow accustomed to the tone-reducing stimuli which may require some acclimatization.

Third appointment: A clinical examination is conducted by PT. Surface gel electrodes are then attached while the participant is instructed in individual muscle activation tests; SENIAM guidelines will be followed for electrode placement and skin preparation, aside from hamstrings and rectus femoris which will follow amended instructions in line with the scientific literature.

GA quality checks the raw electromyography (EMG) signals by visual inspection during the isolated muscle activation tests and during a dynamic trial for movement artefacts, cross-talk, baseline drift and good noise-to-signal ratio.

Reflective markers are then applied in accordance with Plug-in Gait lower body model by PT to collect kinematic and kinetic data.

A resting trial is collected to establish the baseline activity level for each muscle.

The participant is instructed to walk at a self-selected speed along the walkway. Dynamic trials continue until two clean strikes to the middle force plate are collected for the involved leg. Barefoot data is collected first while any additional modifications necessary for electrode placement are made to the ankle-foot orthoses. The order of the orthotic conditions is randomized.

Data will be recorded confidentially using reference codes for participants and stored on a secure server with designated space allocated by the hospital.

ELIGIBILITY:
Inclusion criteria:

* Spastic unilateral cerebral palsy (hemiplegic)
* Use of an ankle-foot orthosis (AFO) during walking because of equinus in the ankle,
* Excessive plantarflexion during walking
* Gross Motor Function Classification System (GMFCS) I or II

Exclusion criteria:

* Orthopedic surgery on the involved lower limb during the previous 12 months
* Treated with BTX-a in muscles of the involved lower limb during the previous 6 months
* Operated with selective dorsal rhizotomy (SDR)
* Passive dorsiflexion in the ankle, passive extension of the knee and hip < 0 degrees (no fixed contractures)

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2017-10-19 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Muscle activity on/off times | 30 minutes
  Linear electromyography profiles of muscle activity (high-pass filtered, rectified and low-pass enveloped) for medial gastrocnemius, tibialis anterior, medial hamstrings, rectus femoris and vastus lateralis during walking. For each condition, gait cycles from two trials will be averaged. Signals will be synchronized to the gait cycle by foot contact/foot off events and normalized to max dynamic peak. On/off times will be defined as a percentage of max dynamic peak.
Median frequency | 30 minutes
  Median frequency [uV] representing firing frequency for each muscle. Averaged for gait cycles from two trials for each condition.
Root-mean-square (RMS) | 30 minutes
  RMS to quantify difference in firing amplitude between conditions; normalized against resting RMS value for same muscle.

SECONDARY OUTCOMES:
Ankle kinematic graph, sagittal plane | 30 minutes
  Average ankle angle [degrees] for each time interval the gait cycle is divided into.
Ankle moment, sagittal plane | 30 minutes
  Average moment [Nm] value for each time interval the gait cycle is divided into.

CONTACTS AND LOCATIONS:
Overall Officials: Ann-Britt Huse, M. Sc., Principal Investigator — Oslo Universety Hospital, Oslo, Norway
Locations (1):
- Oslo University Hospital, Rikshospitalet, Oslo, Norway